CLINICAL TRIAL: NCT06926764
Title: Intertransverse Process Block to Improve Quality of Recovery After Cardiac Surgery With Sternotomy: a Prospective Randomised Controlled Trial
Brief Title: Intertransverse Process Block to Improve Quality of Recovery After Cardiac Surgery With Sternotomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, WONG MAN KIN, Consultant Anaesthesiologist, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ITBP - Acute pain
Record Dates: First submitted 2025-03-25; First posted 2025-04-15 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Acute Postoperative Pain
Keywords: Cardiac surgery; Intertransverse process block; ITPB; CABG; Quality of Recovery; Acute postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional arm (Experimental): Intertransverse process block is performed on patients with injection of 25ml 0.25% levobupivacaine at the retro-SCTL space after a test bolus of 1-2ml 0.9% normal saline. The same procedure is repeated on the other side with same volume of study medication.
  Interventions: Procedure: Intertransverse process block; Drug: Levobupivacaine 0.25%; Device: Ultrasound guided injection with local anaestethic
- Control arm (Sham Comparator): Sham intertransverse process block is performed on patients with injection of 25ml placebo at the retro-SCTL space after a test bolus of 1-2ml 0.9% normal saline. The same procedure is repeated on the other side with same volume of study medication.
  Interventions: Procedure: Sham Block; Drug: Sodium Chloride (NaCl) 0.9 %; Device: Ultrasound guided injection with local anaestethic

INTERVENTIONS:
Procedure: Intertransverse process block — All blocks are performed by an anaesthesiologist who had previously performed ≥50 successful ITPB blocks, using Philips EPIQ ultrasound system, with a curved array transducer (C5-1), and 80mm echogenic nerve block needle. ITPB is performed with the patients positioned in a lateral decubitus position. The target intervertebral level (T4-5) is identified and marked in the preview ultrasound scan. The transducer is placed 2-3 cm lateral to the spinous process. Under strict asepsis, a single-level (T4-5) ultrasound-guided ITPB is performed with the in-plane insertion of the block needle from lateral to medial direction until its tip is at the medial aspect of the retro-SCTL space. After confirming the needle position by distension of the retro-SCTL space after a test bolus injection of 1-2 ml 0.9% normal saline, 25 ml 0.25% levobupivacaine is injected via the nerve block needle in small aliquots. The same procedure is repeated on the other side with the same v
  Arms: Interventional arm
Procedure: Sham Block — All blocks are performed by an anaesthesiologist who had previously performed ≥50 successful ITPB blocks, using Philips EPIQ ultrasound system, with a curved array transducer (C5-1), and 80mm echogenic nerve block needle (SonoTAP; PAJUNK, Germany). ITPB is performed with the patients positioned in a lateral decubitus position. The target intervertebral level (T4-5) is identified and marked in the preview ultrasound scan. The transducer is placed 2-3 cm lateral to the spinous process. Under strict asepsis, a single-level (T4-5) ultrasound-guided ITPB is performed with the in-plane insertion of the block needle from lateral to medial direction until its tip is at the medial aspect of the retro-SCTL space. After confirming the needle position by distension of the retro-SCTL space after a test bolus injection of 1-2 ml 0.9% normal saline, 25 ml placebo is injected via the nerve block needle in small aliquots. The same procedure is repeated on the other side with the same volume study drug.
  Arms: Control arm
Drug: Levobupivacaine 0.25% — Drug used for intertransverse process block (intervention group)
  Arms: Interventional arm
Drug: Sodium Chloride (NaCl) 0.9 % — As placebo for sham block group
  Arms: Control arm
Device: Ultrasound guided injection with local anaestethic — Philips EPIQ ultrasound system, with a curved array transducer (C5-1), and 80mm echogenic nerve block needle (SonoTAP; PAJUNK, Germany)

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy of intertransverse process block (ITPB) in blunting sympathetic response of sternotomy, achieving perioperative opioid-sparing and improving quality of recovery in adult patients undergoing elective cardiac surgery (e.g., coronary artery bypass graft [CABG], valve repair/replacement, or combined CABG/valve procedures).

The main questions it aims to answer are:

1. To investigate the efficacy of intertransverse process block (ITPB) on quality of recovery after cardiac surgery
2. To investigate the efficacy of ITPB on the sympathetic response on incision, intraoperative and postoperative morphine requirement
3. To investigate the efficacy of ITPB on surgical outcomes including time to weaning off mechanical ventilation, length of ICU/ hospital stay and incidence of neuropathic pain after surgery Researchers will compare patients receiving bilateral ITPB with levobupivacaine to those receiving sham blocks to determine if ITPB reduces CPSP, improves pain control, and decreases opioid consumption.

DETAILED DESCRIPTION:
BACKGROUND Acute postoperative pain is common among cardiac surgical patients, particularly within the first 2 days after surgery, with reported at least moderate intensity. Pain is mainly caused by sternotomy incision, surgical dissection, sternal and ribs fracture, injury to intercostal nerves, and also from sites of drainage cannulas and chest tubes. Poorly controlled acute postoperative pain is associated with adverse physiological outcomes that impair the recovery of cardiac surgical patients. It reduced patient satisfaction, delayed postoperative ambulation, and was associated with development of chronic postsurgical pain (CPSP). The association between sternotomy pain and pulmonary complications has been observed, and the sympathetic activation secondary to pain can induce myocardial ischemia and arrhythmias. Pain control has also been pointed out as one of the major concerns to cardiac surgical patients in intensive care unit (ICU).

Opioid-based technique is commonly used in cardiac anaesthesia to blunt the sympathetic response to surgical pain and maintain hemodynamic stability. However, opioids have dose-dependent side effects and excessive use can prolong mechanical ventilation and time spent in intensive care unit. In modern years that fast-track cardiac anaesthesis is being practiced, opioid-sparing techniques and incorporation of regional anaesthesia into cardiac surgical pain management would enable early extubation, mobilization and discharge from ICU. While neuraxial techniques such as spinal and epidural anaesthesia are possible, there are concerns on hemodynamic instability and the potential for neuraxial hematoma after systemic heparinization in cardiac surgery. Thoracic paraspinal blocks such as paravertebral (PVB) and erector spinae plane block (ESPB) seem to be better alternatives to neuraxial techniques. Paravertebral block has more stable hemodynamic profile and was shown to reduce time on mechanical ventilation and improved intraoperative and postoperative opioid consumption. However, there are concerns on pleural puncture and pneumothorax. The close proximity to vascular structures also raise concerns in systemic heparinization in cardiac surgery. ESPB was reported to decrease perioperative morphine consumption and pain score.However, the sensory block was inconsistent. A systematic review reported no difference in postoperative pain intensity. The spread of local anaesthetics in ESPB was unpredictable, resulting in variable anaesthesia and analgesia over anterior hemithorax. Parasternal fascial plane blocks such as superficial and deep parasternal intercostal blocks can avoid the complications associated with neuraxial and paravertebral techniques with favourable outcomes. However, they only cover anterior cutaneous branches of intercostal nerves T2-6 which may not relieve the visceral pain from mediastinum and the pain from chest tubes inserted beyond the dermatomes. Moreover, due to the close proximity of deep parasternal intercostal plane to internal mammary artery (LIMA) and pleura, there are risks of pneumothorax, LIMA injury or hematoma which are considered undesirable in cardiac surgical patients.

Intertransverse process block (ITPB) is a collective name for several reported paraspinal block techniques such as midpoint transverse process block, costotransverse process block or costotransverse foramen block. The nomenclature was standardized through international consensus. ITPB targets paravertebral space by extra-paravertebral injection of local anaesthetics (LA) within the intertransverse tissue complex (ITTC), posterior to the superior costotransverse ligament (SCTL). ITPB anaesthetizes the ventral rami of spinal nerves, the sympathetic trunk, the communicating rami, and demonstrated LA spread into the thoracic paravertebral space with effective analgesia after breast and video-assisted thoracoscopic surgeries. Compared to other regional techniques for pain management in cardiac surgery, ITPB can be technically simpler and safer to avoid pleural puncture, less bleeding concerns in systemic heparinization, yet provides both somatic and visceral analgesia. Randomized controlled trials (RCT) for ITPB in cardiac surgery are sparse. To date, this is the first RCT to evaluate the analgesic efficacy of ITPB in adult cardiac surgical patients. The investigators hypothesized that bilateral ITPB can provide better perioperative analgesia by blunting sympathetic response of sternotomy, achieving perioperative opioid-sparing and improving quality of recovery.

METHODS

Study population and design This is a single-centre, prospective, randomized, double-blinded, placebo-controlled trial at the Prince of Wales Hospital, a university teaching hospital in Hong Kong.

The investigators include adult patients aged 18 or older, undergoing elective coronary artery bypass graft (CABG), valve repair/replacement, or combined CABG/valve procedure via sternotomy. The investigators exclude emergency surgery, redo surgery, history of thoracotomy or mastectomy, patients with history of chronic pain or on chronic opioids or sedatives, renal failure with estimated glomerular filtration rate <30ml/min (calculated by Cockcroft-Gault formula), intraoperative use of remifentanil and unable to provide informed consent.

Randomization and concealment Patients are randomly assigned into two groups by drawing sequentially numbered, coded sealed, opaque envelops each containing the group assignment of either interventional or control group. The sealed envelopes are prepared by a third party who took no further part in the study. The study drug syringes are prepared under strict aseptic techniques by a nurse not involved in the study. ITPB will be performed by a single anaesthesiologist who was blinded to group allocation. The primary care team, blinded to group allocation, performs all surgical procedures using standardized techniques. Anaesthesiologists, nurses and research team, blinded to group allocation, record data intraoperatively, in ICU, and at regular intervals in the cardiac wards.

Ultrasound block placement Patients receive ITPB prior to anaesthesia induction in a lateral decubitus position. All blocks will be done by a single anaesthesiologists who had performed more than 50 successful ITPBs, using a low-frequency curved array transducer (6-1 MHz), and a 80mm echogenic nerve block needle (SonoTAP; PAJUNK, Germany). Ultrasound-guided bilateral ITPB is performed at T4/5 level by counting from cephalad to caudad direction starting from the most prominent spinous process at C7. The transducer is placed transversely to delineate several bony landmarks associated with paravertebral region: the rib, transverse process, inferior articular process and SCLT that are collectively known as the ITTP. Nerve block needle is introduced in-plane and advanced from lateral-to-medical direction until tip is visualized within the retro-SCLT space lateral to the inferior articular process. After negative aspiration of blood, 25ml 0.25% levobupivacaine will be injected on each side in intervention group while sham block with equal volume of normal saline will be injected in the control. During injection, the investigators observe for distension of retro-SCLT space, distension of thoracic paravertebral space and increased echogenicity of SCLT. All patients are tested for anaesthesia (reduced sensation to ice) at bilateral anterior hemithorax 15 minutes after the block. Surgical incision and sternotomy are performed more than 30 minutes after block placement.

Anaesthesia and interventions All patients receive general anaesthesia for the cardiac surgery, which include midazolam 0.01-0.05mg/kg, fentanyl 2-5mcg/kg and rocuronium 0.5-1mg/kg to facilitate intubation with single-lumen cuffed endotracheal tube. Anaesthesia is maintained with sevoflurane and propofol infusion that targeted Bispectral Index 40 to 60. No vasoactive agents are used to lower the blood pressure except fentanyl and morphine that blunt sympathetic response to pain. Administration of opioids will be left to the discretion of the attending anaesthetist. No other analgesics will be used intraoperatively. Patient-controlled analgesia (PCA) morphine is prescribed for 72 hours after operation for postoperative analgesia (1mg bolus, 5 minute lockout time and a safety maximum of 20mg per 4 hour interval). Information about the PCA pump and instructions to use only if the Numeric Rating Scale (NRS) pain score ≥4 will be given to the patient before surgery and repeated in ICU. Oral analgesics including paracetamol 1g and dihydrocodeine 30mg every 6 hours are prescribed by parent surgical team. At the end of the operation, patients are kept sedated with propofol infusion to ICU. It is stopped upon admission to ICU to facilitate weaning from ventilator. Adaptive support ventilation (ASV) is used for weaning. It adjusts the ventilatory parameters depending on lung mechanics and breathing effort.

Data collection Patients are screened the day before operation. Eligible patients are given information sheets regarding the main aspects of the trial and information is discussed with the research nurse before informed consent can be obtained. All data are collected by research team members blinded to group assignment. Patient demographics and body mass index are recorded. Cumulated opioid consumption data and time to first morphine rescue are extracted from PCA pump. At 15 minutes after tracheal extubation and at 2h, 4h, 6h, 8h, 12h, 24h, 48h and 72h post-extubation, pain score at rest and on coughing will be quantified using NRS from 0 to 10. Zero represents no pain at all while 10 points represents the worst pain ever. The patients are asked to rate the overall satisfaction to pain management on a verbal analogue scale (0 = worst possible, 100 = best possible) at the predefined points. The level of sedation is measured using the Ramsay Sedation Scale (1 = anxious, agitated or restless, or both; 2 = co-operative, oriented and tranquil; 3= respond to command only; 4 = exhibit brisk response to light glabellar tap or loud auditory stimulus; 5 = exhibit sluggish response to light glabellar tap or loud auditory stimulus; 6 = exhibits no response). Any nausea and vomiting, and use of rescue antiemetics are documented. The Chinese validated version of the Quality of Recovery Questionnaire (QoR-15) is completed at baseline (preoperatively) and postoperatively at 24 hours and 72 hours after extubation.

Outcome measures Primary outcome is QoR-15 score at 24 and 72 hours after extubation. Secondary outcomes include intraoperative opioid consumption, morphine consumption within 24 and 72 hours after surgery, percentage changes in hemodynamic parameters from baseline within the first 10 minutes of skin incision for sternotomy, postoperative pain score, time of first morphine rescue, patients' satisfaction to pain, time weaned to spontaneous breathing on ASV, time to extubation, side effects from opioids (level of sedation, nausea and vomiting), length of ICU and hospital stay, and neuropathic pain assessment at 3 and 6 months after surgery.

Intraoperative opioids other than morphine are converted into intravenous morphine equivalent dose, and dose of fentanyl used at anaesthesia induction is recorded. Hemodynamic changes following sternotomy are defined as percentage increase in systolic blood pressure (SBP), diastolic blood pressure (DBP), mean arterial pressure (MAP) and heart rate (HR) between the baseline and their peaks within 10 minutes of skin incision for sternotomy. All hemodynamic parameters are automatically recorded using the Anaesthesia Clinical Information System at one-minute interval.

Neuropathic pain at 3 and 6 months after surgery will be assessed using the Douleur Neuropathique en 4 questionnaire (DN4). It is a 10 items questionnaire and the Mandarin Chinese version has been validated in previous study. Each item of DN4 is assigned a score of 0 when the participant answered 'no' and a score of 1 when the participant answered 'yes'. The total DN4 score ranges from 0 to 10, and a score ≥4 indicates a diagnosis of neuropathic pain.

Sample size and statistics Sample size is calculated using G*Power software version 3.1.9.3 (Kiel University, Kiel, Germany) and based on the QoR-15 score at 24 and 72 hours after surgery, which is the primary outcome variable. The minimum clinically important difference (MCID) for the QoR-15 score at 24 hours is 8 and the typical standard deviation (SD) of QoR-15 in the postoperative period ranges between 10-16. Based on these data, for a two-sided test, assuming a type I error of 0.05 and type II error of 0.2, population variance of 144 (SD was assumed to be 12), the investigators calculate a sample size of 36 in each group. Considering a 10% dropout rate, a total of 80 patients (40 patients in each group) will provide 80% power to detect a different in the mean QoR-15 score at 24 hours.

The primary analyses are performed on a modified intention-to-treat basis. Patients are analysed according to their randomized allocated groups but are excluded from the analysis if they do not adhere to the protocol after randomisation. Categorical data is reported as numbers and percentages. Continuous variables are reported as mean (standard deviation) or median (interquartile range) as appropriate after checking for normality using the Shapiro-Wilk's test. Comparison of continuous data is performed by Student's t test and by Mann-Whitney U test for non-normally distributed data. Chi-square test is used to compare groups with categorical variables. Level of significance is set at P<0.05. SPSS 27.0 software (IBM Corp, Armonk, NY) is used for data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged 18 or older
* undergoing elective coronary artery bypass graft (CABG), valve repair/replacement, or combined CABG/valve procedure via sternotomy.

Exclusion Criteria:

* Emergency surgery
* redo surgery
* history of thoracotomy or mastectomy
* patients with history of chronic pain
* patients on chronic opioids or sedatives
* renal failure with estimated glomerular filtration rate <30ml/min (calculated by Cockcroft-Gault formula)
* intraoperative use of remifentanil
* unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
Quality of recovery at 24 hours after extubation | 24 hours after extubation
  Chinese validated version of the Quality of Recovery Questionnaire (QoR-15), range from 0 - 150, with 150 indicating excellent recovery and 0 indicated poor recovery.

SECONDARY OUTCOMES:
Quality of recovery at 72 hours after extubation | 72 hours after extubation
  Chinese validated version of the Quality of Recovery Questionnaire (QoR-15), range from 0 - 150, with 150 indicating excellent recovery and 0 indicated poor recovery.
Intraoperative opioid consumption | Intraoperatively
  Intraoperative opioids other than morphine are converted into intravenous morphine equivalent dose, and dose of fentanyl used at anaesthesia induction is recorded.
Morphine consumption | within 24 and 72 hours after surgery
  Morphine consumption postoperatively
SBP change on incision for sternotomy | within 10 minutes of skin incision of sternotomy
  Systolic blood pressure changes following sternotomy are defined as percentage increase in systolic blood pressure (SBP) between the baseline and their peaks within 10 minutes of skin incision for sternotomy. All hemodynamic parameters are automatically recorded using the Anaesthesia Clinical Information System at one-minute interval.
Postoperative pain score | 15 minutes after tracheal extubation and at 2, 4, 6, 8, 12, 24, 48 and 72 hours post-extubation
  Pain score at rest and on coughing will be quantified using NRS from 0 to 10. Zero represents no pain at all while 10 points represents the worst pain ever.
Time of first rescue morphine | After operation, on average 0 - 3 days after operation, up until first morphine required is recorded if any.
  Time of first rescue morphine required
Patient's satisfaction to pain | 15 minutes after tracheal extubation and at 2, 4, 6, 8, 12, 24, 48 and 72hours post-extubation
  The patients are asked to rate the overall satisfaction to pain management on a verbal analogue scale (0 = worst possible, 100 = best possible) at the predefined points.
Time of weaning to spontaneous ventilation | After operation, on average 0 - 2 days after operation, up until weaning to spontaneous ventilation is recorded.
  At the end of the operation, patients are kept sedated with propofol infusion to ICU. It is stopped upon admission to ICU to facilitate weaning from ventilator. Adaptive support ventilation (ASV) is used for weaning. It adjusts the ventilatory parameters depending on lung mechanics and breathing effort. Time of weaning to spontaneous ventilation is recorded
Time to extubation | Up to 12 hours in ICU
  Time of extubation in postoperative period in ICU
Opioid side effects | 15 minutes after tracheal extubation and at 2, 4, 6, 8, 12, 24, 48 and 72 hours post-extubation
  Including level of sedation measured using the Ramsay Sedation Scale (1 = anxious, agitated or restless, or both; 2 = co-operative, oriented and tranquil; 3= respond to command only; 4 = exhibit brisk response to light glabellar tap or loud auditory stimulus; 5 = exhibit sluggish response to light glabellar tap or loud auditory stimulus; 6 = exhibits no response) and nausea and vomiting andthe use of rescue antiemetics.
Length of stay in ICU and hospital | Up to 30 days after surgery
  Length of stay in ICU and hospital
Postoperative neuropathic pain | 3 months and 6 months after surgery
  Neuropathic pain at 3 and 6 months after surgery will be assessed using the Douleur Neuropathique en 4 questionnaire (DN4). It is a 10 items questionnaire and the Mandarin Chinese version has been validated in previous study. Each item of DN4 is assigned a score of 0 when the participant answered 'no' and a score of 1 when the participant answered 'yes'. The total DN4 score ranges from 0 to 10, and a score ≥4 indicates a diagnosis of neuropathic pain.
DBP changes at incision for sternotomy | within 10 minutes of skin incision of sternotomy
  Diastolic blood pressure changes following sternotomy are defined as percentage increase in diastolic blood pressure (DBP) between the baseline and their peaks within 10 minutes of skin incision for sternotomy. All hemodynamic parameters are automatically recorded using the Anaesthesia Clinical Information System at one-minute interval.
MAP changes at incision for sternotomy | within 10 minutes of skin incision of sternotomy
  Mean arterial blood pressure changes sternotomy are defined as percentage increase in mean arterial blood pressure (MAP) between the baseline and their peaks within 10 minutes of skin incision for sternotomy. All hemodynamic parameters are automatically recorded using the Anaesthesia Clinical Information System at one-minute interval.
HR changes at incision for sternotomy | within 10 minutes of skin incision of sternotomy
  Heart rate changes sternotomy are defined as percentage increase in heart rate between the baseline and their peaks within 10 minutes of skin incision for sternotomy. All hemodynamic parameters are automatically recorded using the Anaesthesia Clinical Information System at one-minute interval.

CONTACTS AND LOCATIONS:
Overall Officials: Henry Wong, Principal Investigator — Hospital Authority

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang H, Qu Z, Miao Y, Zhang Y, Qian L, Hua B, Hua Z. Comparison between ultrasound-guided multi-injection intertransverse process and thoracic paravertebral blocks for major breast cancer surgery: a randomized non-inferiority trial. Reg Anesth Pain Med. 2023 Apr;48(4):161-166. doi: 10.1136/rapm-2022-104003. Epub 2022 Dec 15. PMID 36522043
- [Result] Moorthy A, Ni Eochagain A, Dempsey E, Wall V, Marsh H, Murphy T, Fitzmaurice GJ, Naughton RA, Buggy DJ. Postoperative recovery with continuous erector spinae plane block or video-assisted paravertebral block after minimally invasive thoracic surgery: a prospective, randomised controlled trial. Br J Anaesth. 2023 Jan;130(1):e137-e147. doi: 10.1016/j.bja.2022.07.051. Epub 2022 Sep 13. PMID 36109206
- [Result] Myles PS, Myles DB, Galagher W, Chew C, MacDonald N, Dennis A. Minimal Clinically Important Difference for Three Quality of Recovery Scales. Anesthesiology. 2016 Jul;125(1):39-45. doi: 10.1097/ALN.0000000000001158. PMID 27159009
- [Result] Spallone V, Morganti R, D'Amato C, Greco C, Cacciotti L, Marfia GA. Validation of DN4 as a screening tool for neuropathic pain in painful diabetic polyneuropathy. Diabet Med. 2012 May;29(5):578-85. doi: 10.1111/j.1464-5491.2011.03500.x. PMID 22023377
- [Result] Bouhassira D, Attal N, Alchaar H, Boureau F, Brochet B, Bruxelle J, Cunin G, Fermanian J, Ginies P, Grun-Overdyking A, Jafari-Schluep H, Lanteri-Minet M, Laurent B, Mick G, Serrie A, Valade D, Vicaut E. Comparison of pain syndromes associated with nervous or somatic lesions and development of a new neuropathic pain diagnostic questionnaire (DN4). Pain. 2005 Mar;114(1-2):29-36. doi: 10.1016/j.pain.2004.12.010. Epub 2005 Jan 26. PMID 15733628
- [Result] Wang YF, Yang CC, Ro LS, Tsai YC, Lin KP, Sun WZ, Fang WT, Wang SJ. Development and validation of a Taiwan version of the DN4-T questionnaire. J Chin Med Assoc. 2019 Aug;82(8):623-627. doi: 10.1097/JCMA.0000000000000129. PMID 31169589
- [Result] Bu XS, Zhang J, Zuo YX. Validation of the Chinese Version of the Quality of Recovery-15 Score and Its Comparison with the Post-Operative Quality Recovery Scale. Patient. 2016 Jun;9(3):251-9. doi: 10.1007/s40271-015-0148-6. PMID 26518201
- [Result] Stark PA, Myles PS, Burke JA. Development and psychometric evaluation of a postoperative quality of recovery score: the QoR-15. Anesthesiology. 2013 Jun;118(6):1332-40. doi: 10.1097/ALN.0b013e318289b84b. PMID 23411725
- [Result] Somani S, Makhija N, Chauhan S, Bhoi D, Das S, Bandi SG, Rajashekar P, Bisoi AK. Comparison of Multiple Injection Costotransverse Block and Erector Spinae Plane Block for Post-Sternotomy Pain Relief in Pediatric Patients Undergoing Cardiac Surgery: A Prospective Randomized Comparative Study. J Cardiothorac Vasc Anesth. 2024 Apr;38(4):974-981. doi: 10.1053/j.jvca.2023.12.037. Epub 2023 Dec 29. PMID 38326195
- [Result] Abdelbaser I, Abourezk AR, Badran A, Abdelfattah M. Bilateral Ultrasound-Guided Mid-Point Transverse Process to Pleura Block for Perioperative Analgesia in Pediatric Cardiac Surgery: A Randomized Controlled Study. J Cardiothorac Vasc Anesth. 2023 Sep;37(9):1726-1733. doi: 10.1053/j.jvca.2023.05.021. Epub 2023 May 14. PMID 37296029
- [Result] Karmakar MK, Sivakumar RK, Sheah K, Pangthipampai P, Lonnqvist PA. The Retro Superior Costotransverse Ligament Space as a New Target for Ultrasound-Guided Intertransverse Process Block: A Report of 2 Cases. A A Pract. 2022 Jul 22;16(7):e01610. doi: 10.1213/XAA.0000000000001610. eCollection 2022 Jul 1. PMID 35867848
- [Result] Bhoi D, Narasimhan P, Nethaji R, Talawar P. Ultrasound-Guided Midpoint Transverse Process to Pleura Block in Breast Cancer Surgery: A Case Report. A A Pract. 2019 Feb 1;12(3):73-76. doi: 10.1213/XAA.0000000000000850. PMID 30085935
- [Result] Cho TH, Kwon HJ, O J, Cho J, Kim SH, Yang HM. The pathway of injectate spread during thoracic intertransverse process (ITP) block: Micro-computed tomography findings and anatomical evaluations. J Clin Anesth. 2022 May;77:110646. doi: 10.1016/j.jclinane.2022.110646. Epub 2022 Jan 10. PMID 35021139
- [Result] Costache I, de Neumann L, Ramnanan CJ, Goodwin SL, Pawa A, Abdallah FW, McCartney CJL. The mid-point transverse process to pleura (MTP) block: a new end-point for thoracic paravertebral block. Anaesthesia. 2017 Oct;72(10):1230-1236. doi: 10.1111/anae.14004. Epub 2017 Aug 1. PMID 28762464
- [Result] Bowness JS, Pawa A, Turbitt L, Bellew B, Bedforth N, Burckett-St Laurent D, Delbos A, Elkassabany N, Ferry J, Fox B, French JLH, Grant C, Gupta A, Harrop-Griffiths W, Haslam N, Higham H, Hogg R, Johnston DF, Kearns RJ, Kopp S, Lobo C, McKinlay S, Memtsoudis S, Merjavy P, Moka E, Narayanan M, Narouze S, Noble JA, Phillips D, Rosenblatt M, Sadler A, Sebastian MP, Taylor A, Thottungal A, Valdes-Vilches LF, Volk T, West S, Wolmarans M, Womack J, Macfarlane AJR. International consensus on anatomical structures to identify on ultrasound for the performance of basic blocks in ultrasound-guided regional anesthesia. Reg Anesth Pain Med. 2022 Feb;47(2):106-112. doi: 10.1136/rapm-2021-103004. Epub 2021 Sep 22. PMID 34552005
- [Result] Wong HMK, Chen PY, Tang GCC, Chiu SLC, Mok LYH, Au SSW, Wong RHL. Deep Parasternal Intercostal Plane Block for Intraoperative Pain Control in Cardiac Surgical Patients for Sternotomy: A Prospective Randomized Controlled Trial. J Cardiothorac Vasc Anesth. 2024 Mar;38(3):683-690. doi: 10.1053/j.jvca.2023.11.038. Epub 2023 Nov 30. PMID 38148266
- [Result] Sorenstua M, Zantalis N, Raeder J, Vamnes JS, Leonardsen AL. Spread of local anesthetics after erector spinae plane block: an MRI study in healthy volunteers. Reg Anesth Pain Med. 2023 Feb;48(2):74-79. doi: 10.1136/rapm-2022-104012. Epub 2022 Nov 9. PMID 36351741
- [Result] Oostvogels L, Weibel S, Meissner M, Kranke P, Meyer-Friessem CH, Pogatzki-Zahn E, Schnabel A. Erector spinae plane block for postoperative pain. Cochrane Database Syst Rev. 2024 Feb 12;2(2):CD013763. doi: 10.1002/14651858.CD013763.pub3. PMID 38345071
- [Result] Karmakar MK, Lonnqvist PA. The clinical use of the thoracic erector spinae plane block. Con - ESPB is not useful for thoracic analgesia. J Clin Anesth. 2024 May;93:111353. doi: 10.1016/j.jclinane.2023.111353. Epub 2023 Nov 30. No abstract available. PMID 38039630
- [Result] Dost B, De Cassai A, Balzani E, Tulgar S, Ahiskalioglu A. Effects of ultrasound-guided regional anesthesia in cardiac surgery: a systematic review and network meta-analysis. BMC Anesthesiol. 2022 Dec 29;22(1):409. doi: 10.1186/s12871-022-01952-7. PMID 36581838
- [Result] Macaire P, Ho N, Nguyen T, Nguyen B, Vu V, Quach C, Roques V, Capdevila X. Ultrasound-Guided Continuous Thoracic Erector Spinae Plane Block Within an Enhanced Recovery Program Is Associated with Decreased Opioid Consumption and Improved Patient Postoperative Rehabilitation After Open Cardiac Surgery-A Patient-Matched, Controlled Before-and-After Study. J Cardiothorac Vasc Anesth. 2019 Jun;33(6):1659-1667. doi: 10.1053/j.jvca.2018.11.021. Epub 2018 Nov 19. PMID 30665850
- [Result] Richardson J, Lonnqvist PA, Naja Z. Bilateral thoracic paravertebral block: potential and practice. Br J Anaesth. 2011 Feb;106(2):164-71. doi: 10.1093/bja/aeq378. PMID 21233114
- [Result] Naganuma M, Tokita T, Sato Y, Kasai T, Kudo Y, Suzuki N, Masuda S, Nagaya K. Efficacy of Preoperative Bilateral Thoracic Paravertebral Block in Cardiac Surgery Requiring Full Heparinization: A Propensity-Matched Study. J Cardiothorac Vasc Anesth. 2022 Feb;36(2):477-482. doi: 10.1053/j.jvca.2021.05.001. Epub 2021 May 13. PMID 34099376
- [Result] Capuano P, Sepolvere G, Toscano A, Scimia P, Silvetti S, Tedesco M, Gentili L, Martucci G, Burgio G. Fascial plane blocks for cardiothoracic surgery: a narrative review. J Anesth Analg Crit Care. 2024 Mar 11;4(1):20. doi: 10.1186/s44158-024-00155-5. PMID 38468350
- [Result] Wong WT, Lai VK, Chee YE, Lee A. Fast-track cardiac care for adult cardiac surgical patients. Cochrane Database Syst Rev. 2016 Sep 12;9(9):CD003587. doi: 10.1002/14651858.CD003587.pub3. PMID 27616189
- [Result] Engelman DT, Ben Ali W, Williams JB, Perrault LP, Reddy VS, Arora RC, Roselli EE, Khoynezhad A, Gerdisch M, Levy JH, Lobdell K, Fletcher N, Kirsch M, Nelson G, Engelman RM, Gregory AJ, Boyle EM. Guidelines for Perioperative Care in Cardiac Surgery: Enhanced Recovery After Surgery Society Recommendations. JAMA Surg. 2019 Aug 1;154(8):755-766. doi: 10.1001/jamasurg.2019.1153. PMID 31054241
- [Result] Eisenberg E, Pultorak Y, Pud D, Bar-El Y. Prevalence and characteristics of post coronary artery bypass graft surgery pain (PCP). Pain. 2001 May;92(1-2):11-7. doi: 10.1016/s0304-3959(00)00466-8. PMID 11323122
- [Result] Harrogate SR, Cooper JA, Zawadka M, Anwar S. Seven-year follow-up of persistent postsurgical pain in cardiac surgery patients: A prospective observational study of prevalence and risk factors. Eur J Pain. 2021 Sep;25(8):1829-1838. doi: 10.1002/ejp.1794. Epub 2021 Jun 13. PMID 33982819
- [Result] Roediger L, Larbuisson R, Lamy M. New approaches and old controversies to postoperative pain control following cardiac surgery. Eur J Anaesthesiol. 2006 Jul;23(7):539-50. doi: 10.1017/S0265021506000548. PMID 16677435
- [Result] Puntillo K, Weiss SJ. Pain: its mediators and associated morbidity in critically ill cardiovascular surgical patients. Nurs Res. 1994 Jan-Feb;43(1):31-6. PMID 8295837
- [Result] Lahtinen P, Kokki H, Hynynen M. Pain after cardiac surgery: a prospective cohort study of 1-year incidence and intensity. Anesthesiology. 2006 Oct;105(4):794-800. doi: 10.1097/00000542-200610000-00026. PMID 17006079
- [Result] Gelinas C. Management of pain in cardiac surgery ICU patients: have we improved over time? Intensive Crit Care Nurs. 2007 Oct;23(5):298-303. doi: 10.1016/j.iccn.2007.03.002. Epub 2007 Apr 19. PMID 17448662
- [Result] Milgrom LB, Brooks JA, Qi R, Bunnell K, Wuestfeld S, Beckman D. Pain levels experienced with activities after cardiac surgery. Am J Crit Care. 2004 Mar;13(2):116-25. PMID 15043239
- [Result] Mueller XM, Tinguely F, Tevaearai HT, Revelly JP, Chiolero R, von Segesser LK. Pain location, distribution, and intensity after cardiac surgery. Chest. 2000 Aug;118(2):391-6. doi: 10.1378/chest.118.2.391. PMID 10936130